CLINICAL TRIAL: NCT06268769
Title: Multicentre, Open-label, Randomised, Two-arm, Parallel-group, Superiority Trial to Assess Bioavailability and Practicability of Two Once-daily Tacrolimus Formulations, Envarsus® Compared With Advagraf™, Administered in Kidney Transplant Recipients
Brief Title: Tacrolimus C:D Ratio Measured in Renal Transplant Recipients Treated With Once-daily Prolonged-release Drugs
Acronym: TaC:Drop
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Edward Geissler (Other)
Collaborators: Chiesi Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor-Investigator, Edward Geissler, Head of the Department of Experimental Surgery, University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TaC:Drop; 2023-503531-18-00 (Other: EUCT Number)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Immunosuppression
Keywords: Kidney transplantation; Tacrolimus; Concentration/dose ratio
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: A dynamic allocation technique assigns participants in a 1:1 ratio to one of two treatment arms: Envarsus tablets (test IMP) or Advagraf capsules (comparator IMP). Randomisation is stratified by two factors: a) trial site, in order to minimise systematic treatment bias at the level of the trial centre and reduce the influence of inter-centre variability, and b) participation in the optional pharmacokinetic sub-study, in order to ensure an equal representation of Envarsus- and Advagraf-treated patients in the sub-study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envarsus (Experimental): Participants take prolonged-release tacrolimus tablets (Envarsus) orally once daily and additionally receive standard-of-care immunosuppressive background therapy according to routine practice.
  Interventions: Drug: Tacrolimus Pill
- Advagraf (Active Comparator): Participants take prolonged-release tacrolimus capsules (Advagraf) orally once daily and additionally receive standard-of-care immunosuppressive background therapy according to routine practice.
  Interventions: Drug: Tacrolimus capsule

INTERVENTIONS:
Drug: Tacrolimus Pill — Envarsus tablets dosed to achieve and maintain whole blood trough levels of tacrolimus within a therapeutic range of 5-12 ng/ml during the first 4 weeks post-transplantation, and 5-8 ng/ml thereafter.
  Other Names: Envarsus
  Arms: Envarsus
Drug: Tacrolimus capsule — Advagraf capsules dosed to achieve and maintain whole blood trough levels of tacrolimus within a therapeutic range of 5-12 ng/ml during the first 4 weeks post-transplantation, and 5-8 ng/ml thereafter.
  Other Names: Advagraf
  Arms: Advagraf

SUMMARY:
The goal of this clinical trial is to compare the bioavailability and practicability of two different formulations of tacrolimus in kidney transplant recipients. The main objective is to demonstrate that Envarsus® (test drug) has superior (higher) oral bioavailability compared with Advagraf™ (comparator drug) at 12 weeks after kidney transplantation. The trial also aims to compare the practicability (handling) of the two drugs using a series of pharmacokinetic parameters and to explore the relationship between drug bioavailability and long-term clinical outcomes, with a special focus on dose-dependent adverse reactions, measured until 3 years post-transplantation. The trial incorporates a pharmacokinetic sub-study designed to profile the peak tacrolimus blood concentration up to 6 hours after drug intake on the day of the 12-week study visit.

DETAILED DESCRIPTION:
This clinical trial aims to compare the bioavailability and practicability of two alternative once-daily formulations of tacrolimus in patients who have received either a first or second kidney transplant and require prophylactic immunosuppressive treatment to prevent allograft rejection. Trial participants are randomised within 7 days prior to kidney transplantation surgery in a 1:1 ratio to two alternative treatment arms containing either Envarsus (test arm) or Advagraf (comparator arm) as first-line calcineurin inhibitor within a standard-of-care immunosuppressive regimen. Tacrolimus blood trough levels and drug doses are monitored at regular intervals to measure a dose-normalised trough level (concentration/dose, C/D ratio) as an estimate of tacrolimus bioavailability.

The primary objective is to demonstrate that the C/D ratio of tacrolimus measured in kidney transplant recipients treated with Envarsus® (test drug) is superior to (higher than) the C/D ratio measured in patients treated with Advagraf™ (comparator drug) at 12 weeks post-transplantation. The trial also aims to compare the practicability (handling) of these two once-daily drug formulations using a series of pharmacokinetic parameters that will measure the speed with which therapeutic blood trough levels are attained and the ease with which stable blood trough levels are maintained over time.

Secondarily, TaC:Drop aims to explore the relationship between the early C/D ratio measured at 12 weeks post-transplantation and later clinical outcomes measured until three years post-transplantation. The study aims to investigate whether a superior pharmacokinetic drug profile is associated with fewer and milder dose-dependent drug toxicities and superior kidney graft function, as measured by long-term safety and efficacy parameters.

Drug pharmacokinetics will be explored in greater detail during a sub-study designed to profile the peak blood concentration of Envarsus® and Advagraf™ at 12 weeks post-transplantation in patients who volunteer to provide three additional blood samples at two-hour intervals after drug intake on the day of the 12-week trial visit. Participation in this sub-study is voluntary and available to all trial centres and all trial patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Adult (≥18 years old) male or female
3. Renal insufficiency necessitating kidney transplantation and approved to receive a first or second kidney allograft from a living or deceased organ donor
4. ABO blood type compatible with the donor kidney
5. Able to swallow an oral formulation of tacrolimus in tablet or capsule form

Exclusion Criteria:

1. Multi-organ transplantation
2. Any previous solid organ transplantation (other than a first kidney allograft)
3. For recipients of a second kidney transplant: loss of first kidney transplant within 2 years after transplantation owing to immunological reasons or recurrence of the underlying renal disease
4. Patient and/or donor is positive for HCV, HBV or HIV
5. History of any malignancy that could not be curatively treated
6. Ongoing abuse of drugs or alcohol
7. Signs of advanced liver disease or any signs of liver decompensation
8. Ongoing uncontrolled systemic infection
9. Severe diarrhoea, vomiting, active peptic ulcer, previous bariatric surgery, or any other gastrointestinal disorder that may affect absorption of tacrolimus
10. Planned or foreseeable use of cyclosporine, belatacept or any tacrolimus preparation other than Envarsus® or Advagraf™
11. Known contraindication or hypersensitivity to tacrolimus, and/or to any of the excipients listed in section 6.1 of the Summary of Product Characteristics (SmPC) of both Envarsus® and Advagraf™, and/or to any other macrolides
12. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
13. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless using a highly-effective method of contraception
14. Participation in another interventional clinical trial in the time period starting from 4 weeks prior to randomisation and throughout the entire trial period
15. Any condition or factor which, in the judgement of the investigator, would place the subject at undue risk, invalidate communication with the investigator or study team, or hamper compliance with the trial protocol or follow-up schedule
16. Inability to freely give informed consent (e.g. individuals under legal guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Dose-normalised blood trough level of tacrolimus (concentration/dose ratio) | 12 weeks after kidney transplantation
  To calculate C/D ratio, "concentration" is the blood trough level of tacrolimus measured in a blood sample collected immediately prior to drug dosing on the day of the 12-week trial visit and "dose" is the daily dose taken by the patient on the day prior to the visit. C/D ratio is measured as a surrogate for tacrolimus bioavailability (i.e. systemic exposure per mg of drug). The primary endpoint uses a blood trough level reading that is measured in a central laboratory.

SECONDARY OUTCOMES:
Time to reach the first trough level in target range | Time period measured in days, assessed within the first 2 weeks after kidney transplantation
  Reaching the target range is defined as two consecutive readings within the initial target range of 5-12 ng/ml; time is measured to the date of the first in-range reading
Proportion of patients with trough levels lower, within, or higher than the target range | 4 days, 14 days, 28 days and 12 weeks after kidney transplantation
Mean tacrolimus trough level and inter-patient variability (range) of tacrolimus trough levels | 4 days, 14 days, 28 days and 12 weeks after kidney transplantation
Mean daily dose of tacrolimus and inter-patient variability (range) of tacrolimus daily dose | 4 days, 14 days, 28 days and 12 weeks after kidney transplantation
Tacrolimus concentration/dose (C/D) ratio | 4 days, 14 days, 28 days and 1, 2, 3 years after kidney transplantation
  The secondary endpoint using C/D ratio data takes a blood trough level reading that is measured in the local laboratory at the trial site.
Intra-patient variability of C/D ratio and daily dose | Measured over the time points: day 4, day 14, day 28 and week 12
Treatment failure rate | 12 weeks and 1, 2, 3 years after kidney transplantation
  A composite endpoint of biopsy-proven acute rejection, graft failure (defined as initiation of renal dialysis or re-transplantation), or death (from any cause)
Time to treatment failure after transplantation | Measured until 3 years after kidney transplantation
  Treatment failure is a composite endpoint of biopsy-proven acute rejection, graft failure (defined as initiation of renal dialysis or pre-emptive re-transplantation), or death (from any cause)
Incidence rate, severity and time to clinically-confirmed biopsy-proven acute rejection | 12 weeks and 1, 2, 3 years after kidney transplantation
  Clinically-confirmed biopsy-proven acute rejection requires both a clinical diagnosis of rejection by an investigator and a histopathological diagnosis of rejection in a for-cause biopsy. Subclinical rejection diagnosed in a protocol biopsy is therefore excluded from this definition.
Incidence rate of graft failure | 12 weeks and 1, 2, 3 years after kidney transplantation
  Graft failure is defined as initiation of renal dialysis or pre-emptive re-transplantation
Mortality rate | 12 weeks and 1, 2, 3 years after kidney transplantation
  Mortality rate measures death from any cause
Graft function measured by eGFR (estimated glomerular filtration rate) | 4 days, 14 days, 28 days, 12 weeks and 1, 2, 3 years after kidney transplantation
  eGFR calculated according to the CKD-EPI formula
Incidence rate of for-cause biopsies | 12 weeks after kidney transplantation
Incidence rate of acute rejection episodes requiring treatment | 12 weeks after kidney transplantation
Incidence rate of steroid-resistant episodes of biopsy-proven acute rejection | 12 weeks and 1 year after kidney transplantation
Incidence rate of delayed graft function | Measurable within the first 2 weeks after kidney transplantation
  Delayed graft function is defined as the need for more than one episode of dialysis after transplantation
Incidence rate of primary non-function of the renal allograft | Measurable within the first 12 weeks after kidney transplantation
  Primary non-function is defined as the necessity for ongoing chronic dialysis
Incidence of hepatotoxicity | 12 weeks and 1, 2, 3 years after kidney transplantation
  Hepatotoxicity is defined as GPT or GOT levels ≥ 2.5 x upper limit of normal range
Incidence of CMV and BKV infection (including organ manifestation, if relevant) | 12 weeks and 1 year after kidney transplantation
Incidence, type, severity and seriousness of adverse reactions (ARs) | 12 weeks and 3 years after kidney transplantation
Blood pressure | 12 weeks and 1, 2, 3 years after kidney transplantation
Incidence of de novo tremor | 12 weeks and 3 years after kidney transplantation
  Incidence and severity of tremor based on medical assessment by the investigator
Incidence of gastrointestinal disorders requiring diagnostic investigation | 12 weeks and 3 years after kidney transplantation
Incidence of new onset diabetes mellitus after transplantation (NODAT) | 12 weeks and 1, 2, 3 years after kidney transplantation
  NODAT is defined as HbA1c ≥ 6.5% or 47.5 mmol/mol or fasting plasma glucose ≥ 126 mg/dl on two separate occasions
Recurrence of primary kidney disease | 12 weeks and 3 years after kidney transplantation
Incidence of de novo DSA | Detected within the first year after kidney transplantation
Patient-reported health-related quality-of-life measured using the Kidney Transplant Questionnaire-34 (KTQ-34) | 12 weeks and 3 years after kidney transplantation
  The KTQ-34 is a renal transplantation-specific instrument that measures quality-of-life in five dimensions. It is a self-administered questionnaire that is completed in writing by the trial patients.
Doses and duration of glucocorticosteroid treatment | 12 weeks and 1, 2, 3 years after kidney transplantation
Dose of mycophenolate | 12 weeks and 1, 2, 3 years after kidney transplantation
  Including both mycophenolate mofetil and mycophenolic acid
Incidence and time to study treatment discontinuation | 3 years after kidney transplantation
Incidence, time to and reason for patient withdrawal from study | 3 years after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Banas, MD, Principal Investigator — University Hospital Regensburg
Locations (9):
- Germany (9):
  - University Hospital Aachen, Department of General, Visceral and Transplant Surgery, Aachen
  - Charité Universitätsmedizin, Department of Nephrology and Medical Intensive Care, Berlin
  - University Hospital Dresden, Division of Nephrology, Dresden
  - University Medical Center Hamburg-Eppendorf, Internal Medicine III (Nephrology, Rheumatology, Endocrinology), Hamburg
  - Hannover Medical School, Department of General, Visceral and Transplant Surgery, Hanover
  - University Hospital Jena, Internal Medicine III, Nephrology, Jena
  - University Medical Center of the Johannes Gutenberg University Mainz, Medical Clinic I. (Nephrology), Mainz
  - University Hospital Münster, Medical Clinic D, Münster
  - University Hospital Regensburg, Department of Nephrology, Regensburg

IPD SHARING:
Plan to Share IPD: No